CLINICAL TRIAL: NCT06696144
Title: Carriage of Resistant Bacteria on Surfaces and Staff in a Complex Nursing Unit for Patients with Resistant Bacteria
Brief Title: Testing Carriage of Resistant Bacteria Using Swabs on Surfaces and Staff in a Complex Nursing Unit for Patients with Resistant Bacteria
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shmuel Harofeh Hospital, Geriatric Medical Center (Other Government)
Responsible Party: Principal Investigator, Yochai Levy, Hospital deputy director, Shmuel Harofeh Hospital, Geriatric Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SH-109-23
Record Dates: First submitted 2024-11-04; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Multi Drug Resistant Department; Multi Drug Resistant Bacteria
Keywords: MDR, VRE, CRE, older adults, long term care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Skin swabs for multi drug resistant bacteria — Swabs from personal items or skin will be obtained from stuff and analyzed to detect CVE or VRE bacteria using Automated Susceptibility Testing

SUMMARY:
Impact of Care Team and Surfaces on the Spread of Resistant Bacteria in a Specialized Complex Nursing Unit for MDR Pathogen Carriers

Background Multi-drug resistant (MDR) bacteria present a severe clinical and epidemiological challenge, typically managed through strict isolation and continuous monitoring. Transmission patterns among long-term care patients remain unclear. At "Shmuel Harofe" Geriatric Hospital, a dedicated MDR skilled care department was established to reduce infection risks in other hospital settings. It's uncertain if patients in this dedicated unit are more exposed to new bacterial colonizations. Contamination may stem from surfaces in rooms or shared spaces, or from the care team.

Research Objectives

1. To assess whether care team members working in MDR units serve as vectors for infection via skin carriage or personal items.
2. Analyze the presence of resistant bacteria on surfaces in both private and shared spaces within the unit to understand infection transmission risks.

Hypotheses

1. The MDR unit care team does not broadly carry resistant pathogens on their skin or items and does not significantly transmit infections.
2. Surface contamination will be mostly confined to patient rooms, with limited cases on shared surfaces.

Study Design Comparative cross-sectional study with a retrospective cohort component.

Study Population

1. Care Team: All staff in Shmuel Harofe's MDR department (doctors, nursing staff, medical, sanitary, and cleaning staff).
2. Surfaces in Departments: Surfaces in MDR patients' rooms and shared areas in the dedicated MDR unit. Surfeces will be revised acording to a test sampels.

Methods and Materials

1. Staff Sampling: Swabs for CRE and VRE carriage will be collected from hands, facial skin, bags, shoes, cell phones, glasses, and ID badges at the start and end of shifts in the MDR unit.
2. Surface Sampling: Samples from patient environments (e.g., bed railings, cabinets, light switches) and shared areas (e.g., dining tables, door handles, keyboards, and public phones).
3. Clinical Data Collection: Epidemiological data (age, gender, functional status, medical background, length of stay) for statistical analysis.

Statistical Analysis:

* Comparative analysis of bacterial carriage among staff in the MDR unit versus similar wards.
* Analysis of bacterial carriage frequency on surfaces in the MDR unit versus other wards using logistic regression models to assess the relationship between surface type and contamination levels.

Ethics Informed consent will be obtained from staff for sample collection, with data anonymity preserved.

Potential Contributions The study aims to clarify the roles of care staff and surfaces in transmitting resistant bacteria in dedicated units. Insights into transmission mechanisms may aid in developing improved protocols for patient and staff protection and provide recommendations for hygiene and control procedures in healthcare settings.

ELIGIBILITY:
Inclusion Criteria: Works in the hospitals MDR department -

Exclusion Criteria: Non

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of positive swabs for CRE and VRE bacteria in care team members working in MDR units. | 3 month
  Several swabs for VRE and CRE bacteria will be taken from personal items and skin from staff working in a MDR department to access if they serve as vectors for infection via skin carriage or personal items.

IPD SHARING:
Plan to Share IPD: No